CLINICAL TRIAL: NCT01619059
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Triple Therapy With Saxagliptin Added to Dapagliflozin in Combination With Metformin Compared to Therapy With Placebo Added to Dapagliflozin in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin and Dapagliflozin
Brief Title: Safety and Efficacy of Saxagliptin in Triple Therapy to Treat Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CV181-168; 2011-006323-37 (EudraCT Number)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Saxagliptin+Dapagliflozin+Metformin IR (Experimental)
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin; Drug: Metformin IR
- Arm 2: Placebo+Dapagliflozin+Metformin IR (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Metformin IR; Drug: Placebo matching with Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 5 mg, Once daily, Up to 52 weeks
  Other Names: Onglyza
  Arms: Arm 1: Saxagliptin+Dapagliflozin+Metformin IR
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Once daily, Up to 52 weeks
Drug: Metformin IR — Tablets, Oral, ≥ 1500mg, Twice daily, Up to 52 weeks
Drug: Placebo matching with Saxagliptin — Tablets, Oral, 0 mg, Once daily, Up to 52 weeks
  Arms: Arm 2: Placebo+Dapagliflozin+Metformin IR

SUMMARY:
The purpose of this study is to learn if BMS-477118 (Saxagliptin) as part of a triple combination therapy can improve (decrease) hemoglobin A1c in patients with type 2 diabetes after 24 weeks of treatment compared to a 2 drug oral antidiabetic therapy. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria

1. Signed Written Informed Consent

   a) Subjects must be willing and able to give signed and dated written informed consent.
2. Target Population

   1. Subjects with T2DM with inadequate glycemic control, defined as central laboratory HbA1c ≥ 8.0 and ≤ 11.5% obtained at the screening visit (ie Week -18 visit)
   2. Stable metformin therapy for at least 8 weeks prior to screening visit at a dose ≥ 1500 mg per day.
   3. C-peptide ≥ 1.0 ng/mL (0.34 nmol/L) at screening visit.
   4. BMI ≤ 45.0 kg/m2 at the screening visit.
3. Age and Reproductive Status

   1. Men and women, aged ≥ 18 years old at time of screening visit.
   2. Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. See Section 3.3.3 for the definition of WOCBP.
   3. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
   4. Women must not be breastfeeding
   5. Sexually active fertile men must use effective birth control if their partners are WOCBP.

Exclusion Criteria

1. Target Disease Exceptions

   1. History of diabetes insipidus
   2. Symptoms of poorly controlled diabetes that would preclude participation in this trial including but not limited to marked polyuria and polydipsia with greater than 10% weight loss during the three months prior to screening, or other signs and symptoms.
   3. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
2. Medical History and Concurrent Diseases

   1. History of bariatric surgery or lap-band procedure within 12 months prior to screening.
   2. Any unstable endocrine, psychiatric or rheumatic disorders as judged by the Investigator.
   3. Subject who, in the judgment of the investigator, may be at risk for dehydration or volume depletion that may affect the interpretation of efficacy or safety data and concomitant use of loop diuretics in countries where this is not recommended as per the Dapagliflozin label.
   4. Subject is currently abusing alcohol or other drugs or has done so within the last 6 months.

      Acute Vascular Event:
   5. Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg.

      Note: Subjects with SBP ≥ 160mmHg and < 180mmHg or a DBP ≥ 100 mmHg and < 110mmHg will be able to enter the lead-in period, provided their hypertension treatment is adjusted as deemed appropriate by the investigator. These subjects cannot be randomized if their blood pressure remains with SBP ≥ 160 mmHg or DBP ≥ 100 mmHg measured at Day 1.
   6. Cardiovascular Disease within 3 months of the screening visit [ie myocardial infarction, cardiac surgery or revascularization (CABG/PTCA), unstable angina, stroke or transient ischemic attack (TIA)].
   7. Congestive heart failure as New York Association (NYHA) class IV (see Appendix 1), unstable or acute congestive heart failure. Note: eligible patients with congestive heart failure, especially those who are on diuretic therapy, should have careful monitoring of their volumes status throughout the study.

      Renal Diseases:
   8. Moderate or severe impairment of renal function [defined as eGFR < 60 mL/min/1.73 m2 (estimated by MDRD) or serum creatinine (Scr) ≥ 1.5 mg/dL in males or ≥ 1.4 mg/dL in females.]
   9. Conditions of congenital renal glucosuria

      Hepatic Diseases:
   10. Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic insufficiency, including subjects with ALT and/or AST > 3x ULN and or Total Bilirubin > 2.5 x ULN.

       Hematological and Oncological Disease/Conditions
   11. History of hemoglobinopathy, with the exception of sickle cell trait (SA) or thalassemia minor; or chronic or recurrent hemolysis.
   12. Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma)
   13. Known immunocompromised status, including but not limited to, individuals who have undergone organ transplantation or who are positive for the human immunodeficiency virus.
   14. Donation of blood or blood products to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 6 months prior to the screening visit.

       Prohibited treatment and therapies
   15. Administration of any antihyperglycemic therapy, other than metformin, for more than 14 days (consecutive or not) during the 12 weeks prior to screening, as well as previous participation in any DPP-4 or SGLT-2 inhibitor trial is an exclusion criterion.
   16. Current treatment with potent cytochrome P450 3A4/5 inhibitors (in countries where dose adjustment would be required by the saxagliptin label).
   17. Administration of any other investigational drug or participation in any interventional clinical studies within 30 days of planned screening to this study. Subjects who failed to satisfy all eligibility criteria at screening and did not enter the lead-in or open-label period in CV181-169 or MB102-129 studies specifically, do not need to wait 30 days.
3. Physical and Laboratory Test Findings

   1. Hemoglobin ≤ 11.0 g/dL (110 g/L) for men; hemoglobin ≤ 10.0 g/dL (100 g/L) for women
   2. Male subjects with microscopic hematuria present at Week -18 or Week -16 AND no common cause that can be confirmed. Male subjects with a confirmed common cause can be entered into the open-label phase with a documented negative result for hematuria microscopic urinalysis performed by the central laboratory.

      NOTE: Female subjects with hematuria can be entered into the open-label phase and be randomized, but should be investigated according to local standards and best clinical practices. (See Appendix 3)
   3. Other central laboratory test findings:

      * Abnormal free T4 values. Abnormal thyroid stimulating hormone (TSH) value at screening will be further evaluated by free T4. Subjects with abnormal free T4 values will be excluded.
      * Positive for hepatitis B surface antigen
      * Positive for anti-hepatitis C virus antibody
4. Allergies and Adverse Drug Reaction

   a) Subjects who have contraindications to therapy as outlined in the saxagliptin and dapagliflozin Investigator Brochure, the local saxagliptin or dapagliflozin package insert or the local metformin package insert, including current treatment with potent cytochrome P450 3A4/5 inhibitors (in countries where dose adjustment would be required by the local saxagliptin label).
5. Sex and Reproductive Status

   a) Women who are pregnant
6. Other Exclusion Criteria

   1. Prisoners or subjects who are involuntarily incarcerated.
   2. Subject who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (74):
- United States (34):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Terence T. Hart, Md, Muscle Shoals, Alabama
  - Mesa Family Medical Center, Mesa, Arizona
  - Clinical Research Advantage Inc/Desert Clinical Research Llc, Mesa, Arizona
  - Clinical Research Advantage, Inc, Phoenix, Arizona
  - Clinical Research Advantage, Inc./ Stonecreek Medical Associates, Pc, Phoenix, Arizona
  - Beach Physicians Clinical Research Corp., Huntington Beach, California
  - Torrance Clinical Research, Lomita, California
  - Randall G. Shue, Do, Inc., Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Cassidy Medical Group/Clinical Research Advantage, Vista, California
  - Infosphere Clinical Research, Inc., West Hills, California
  - New West Physicians, Pc, Golden, Colorado
  - Southeast Clinical Research, Llc, Chiefland, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Medical Research Unlimited, Llc, Hialeah, Florida
  - University Of Florida Endocrinology & Diabetes, Jacksonville, Florida
  - Care Partners Clinical Research, Llc, Jacksonville, Florida
  - Clinical Research Of Miami, Inc., Miami, Florida
  - Clinical Research Advantage, Inc., Evansville, Indiana
  - Clinical Research Advantage, Evansville, Indiana
  - Mercy Health Research, St Louis, Missouri
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - Joslin Diabetes Center Affiliate Of Snhmc, Nashua, New Hampshire
  - N. Shore Diabetes & Endoc Assoc, New Hyde Park, New York
  - Digiovanna Institute For Medical Education & Research, North Massapequa, New York
  - Barat Research Group, Inc., Charlotte, North Carolina
  - Sterling Research Grp, Ltd., Cincinnati, Ohio
  - Physicians Research, Inc., Zanesville, Ohio
  - Tlm Medical Services, Columbia, South Carolina
  - Family Medicine Of Sayebrook, Myrtle Beach, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Vanderbilt Diabetes Center, Nashville, Tennessee
  - Padre Coast Clinical Research, Corpus Christi, Texas
- Canada (7):
  - Local Institution, Moncton, New Brunswick
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Brampton, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Czechia (3):
  - Local Institution, Hradec Králové
  - Local Institution, Karlovy Vary
  - Local Institution, Prague
- Hungary (4):
  - Local Institution, Balatonfüred
  - Local Institution, Budaörs
  - Local Institution, Budapest
  - Local Institution, Zalaegerszeg
- Mexico (5):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Del. Benito Juarez
  - Local Institution, Veracruz
- Poland (9):
  - Local Institution, Bialystok
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Pszczyna
  - Local Institution, Puławy
  - Local Institution, Szczecin
  - Local Institution, Warsaw
  - Local Institution, Węgrów
  - Local Institution, Wroclaw
- Research & Cardiovascular Corp, Ponce, Puerto Rico
- Romania (7):
  - Local Institution, Brasov, Brașov County
  - Local Institution, Bucharest, Bucharest
  - Local Institution, Bucharest
  - Local Institution, Constanța
  - Local Institution, Craiova
  - Local Institution, Galati
  - Local Institution, Ploieşti
- Russia (4):
  - Local Institution, Kursk
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Yaroslaval

REFERENCES:
- [Derived] Mathieu C, Catrinoiu D, Ranetti AE, Johnsson E, Hansen L, Chen H, Garcia-Sanchez R, Iqbal N, Celinski A. Characterization of the Open-Label Lead-In Period of Two Randomized Controlled Phase 3 Trials Evaluating Dapagliflozin, Saxagliptin, and Metformin in Type 2 Diabetes. Diabetes Ther. 2018 Aug;9(4):1703-1711. doi: 10.1007/s13300-018-0445-x. Epub 2018 May 25. PMID 29802530
- [Derived] Matthaei S, Catrinoiu D, Celinski A, Ekholm E, Cook W, Hirshberg B, Chen H, Iqbal N, Hansen L. Randomized, Double-Blind Trial of Triple Therapy With Saxagliptin Add-on to Dapagliflozin Plus Metformin in Patients With Type 2 Diabetes. Diabetes Care. 2015 Nov;38(11):2018-24. doi: 10.2337/dc15-0811. Epub 2015 Aug 31. PMID 26324329
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 315 participants randomized, 298 completed Short-Term (ST) treatment period. Of 297 participants entered Long-Term (LT) treatment period, 280 completed.
Groups:
- Placebo + Dapagliflozin 10mg + Metformin: Participants received Saxagliptin-matching placebo, dapagliflozin 10mg once daily plus open-label metformin for up to 52 weeks
- Saxagliptin 5mg + Dapagliflozin 10mg + Metformin: Participants received Saxagliptin 5mg, dapagliflozin 10mg once daily plus open-label metformin for up to 52 weeks
Period: Short-Term (ST) Treatment Period
Arm/Group | Placebo + Dapagliflozin 10mg + Metformin | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin
Started | 162 | 153
Completed | 156 | 142
Not Completed | 6 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Non-compliance, not Met Study Criteria | 1 | 2
Period: Long-Term (LT) Treatment Period
Arm/Group | Placebo + Dapagliflozin 10mg + Metformin | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin
Started | 155 | 142
Completed | 147 | 133
Not Completed | 8 | 9
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Not Met Study Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Dapagliflozin 10mg + Metformin | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin | Total
Number analyzed (Participants) | 162 | 153 | 315
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 54.5 (9.32) [27 to 78] | 54.7 (9.83) [27 to 77] | 54.6 (9.56) [27 to 78]
Age, Customized [Number; unit: Participants]
  < 65 | 140 | 132 | 272
  >= 65 | 22 | 21 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 80 | 166
  Male | 76 | 73 | 149
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN/ALASKA NATIVE | 2 | 0 | 2
  ASIAN | 8 | 5 | 13
  BLACK/AFRICAN AMERICAN | 9 | 11 | 20
  OTHER | 2 | 1 | 3
  WHITE | 141 | 136 | 277

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained at Week 24 in the double-blind period, including observations prior to rescue.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24
Measure: Mean (Standard Error); unit: Percent of glycosylated haemoglobin
Arm/Group | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin | Placebo + Dapagliflozin 10mg + Metformin
Number analyzed (Participants) | 139 | 149
Percent of glycosylated haemoglobin | -0.51 (0.0624) | -0.16 (0.0605)
Statistical Analysis 1: Comparison: Saxagliptin 5mg + Dapagliflozin 10mg + Metformin vs Placebo + Dapagliflozin 10mg + Metformin; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Tested at alpha=0.05; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.52 to -0.18], Standard Error of Mean 0.0870

2. Secondary Outcome: Adjusted Mean Change From Baseline in 2-hour Post Prandial Glucose (PPG) From a Liquid Meal Tolerance Test (MTT) at Week 24
Description: Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. PPG measurements were obtained at Week 24 in the double-blind period, including observations prior to rescue.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing PPG values at baseline and Week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin | Placebo + Dapagliflozin 10mg + Metformin
Number analyzed (Participants) | 135 | 144
mg/dL | -37.1 (3.286) | -31.3 (3.182)
Statistical Analysis 1: Comparison: Saxagliptin 5mg + Dapagliflozin 10mg + Metformin vs Placebo + Dapagliflozin 10mg + Metformin; Test type: Superiority or Other; p = 0.2014, Mixed Models Analysis — Secondary endpoints were tested at alpha=0.05, applying the hierarchical order for the sequential testing procedure; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-14.9 to 3.1], Standard Error of Mean 4.576

3. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose at Week 24
Description: Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained at Week 24 in the double-blind period, including observations prior to rescue.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing FPG values at baseline and Week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin | Placebo + Dapagliflozin 10mg + Metformin
Number analyzed (Participants) | 139 | 146
mg/dL | -9.1 (2.644) | -5.3 (2.590)
Statistical Analysis 1: Comparison: Saxagliptin 5mg + Dapagliflozin 10mg + Metformin vs Placebo + Dapagliflozin 10mg + Metformin; Test type: Superiority or Other; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-11.0 to 3.6], Standard Error of Mean 3.713

4. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and were not missing baseline and Week 24 (LOCF) values
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin | Placebo + Dapagliflozin 10mg + Metformin
Number analyzed (Participants) | 139 | 146
Percent of participants | 35.3 (2.644) [28.2 to 42.4] | 23.1 (2.590) [16.9 to 29.3]
Statistical Analysis 1: Comparison: Saxagliptin 5mg + Dapagliflozin 10mg + Metformin vs Placebo + Dapagliflozin 10mg + Metformin; Test type: Superiority or Other; Risk Difference (RD) = 12.2, 95% CI 2-sided [3.4 to 21.0], Standard Error of Mean 4.504

ADVERSE EVENTS:
Arm/Group | Placebo + Dapagliflozin 10mg + Metformin | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin
Serious Adverse Events (participants affected / at risk) | 11/162 | 7/153
Other Adverse Events (participants affected / at risk) | 37/162 | 37/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Dapagliflozin 10mg + Metformin (N=162) | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin (N=153)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
HERNIA (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Dapagliflozin 10mg + Metformin (N=162) | Saxagliptin 5mg + Dapagliflozin 10mg + Metformin (N=153)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 8 (8)
NASOPHARYNGITIS (Infections and infestations) | 8 (8) | 9 (10)
URINARY TRACT INFECTION (Infections and infestations) | 11 (13) | 11 (16)
HEADACHE (Nervous system disorders) | 12 (13) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No